CLINICAL TRIAL: NCT01605201
Title: Tissue Engineered Nasal Cartilage for Regeneration of Articular Cartilage in the Knee After Traumatic Injury - a Phase I Clinical Trial-
Brief Title: Tissue Engineered Nasal Cartilage for Regeneration of Articular Cartilage
Acronym: Nose2Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Deutsche Arthrose-Hilfe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92/11; TpP-I-2012-001 (Other: Swissmedic)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Cartilage Lesion; Degenerative Lesion of Articular Cartilage of Knee
Keywords: Chondral lesions in the knee after traumatic injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implantation of cartilage graft (Experimental)
  Interventions: Biological: Tissue engineered cartilage graft

INTERVENTIONS:
Biological: Tissue engineered cartilage graft — Autologous nasal chondrocytes expanded in vitro and cultured in a collagen type I//III scaffold

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of implanting an engineered cartilage graft obtained by culturing expanded autologous nasal chondrocytes within a collagen type I/III membrane into the cartilage defect on the femoral condyle and/or trochlea of the knee after a traumatic injury.

DETAILED DESCRIPTION:
Articular cartilage injuries are a prime target for regenerative techniques, since spontaneous healing is poor and untreated defects predispose to osteoarthritis. Common current strategies such as arthroscopic debridement, microfracture, autologous osteochondral grafting, use of allografts and autologous chondrocytes implantation (ACI) still have drawbacks such as long and complex rehabilitation times, technically challenging operation techniques, defect-size limitations, donor-site morbidity, limited graft material and high costs. Furthermore many techniques show unsatisfactory long term results due to inferior quality of repair tissue as compared to native cartilage or have yet to prove the cost versus benefit. These drawbacks could be overcome by using a tissue engineered nasal cartilage graft, thereby reducing donor site morbidity without introducing additional risk of complication or technically challenging techniques.

This study is a phase I, prospective, uncontrolled, investigator initiated clinical trial involving 25 patients, with the objective of demonstrating safety and feasibility in the use of engineered nasal cartilage grafts for repair of articular cartilage. The specific surgical target of the trial is the repair of one or two full-thickness cartilage defects from 2 cm2 to 8 cm2 (per lesion, not exceeding a total of 8 cm2 for all lesions) due to traumatic injury on the femoral condyle and/or trochlea of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Size of the defect on the femoral cartilage:one or two symptomatic lesion(s) grade III-IV from 2 cm2 to 8 cm2 at the femoral condyle and/or trochlea
* Other:
* Age: 18-55 years
* Written informed consent by the patient

Exclusion Criteria:

* Defect:

  * Lesions smaller than 2cm2 or greater than 8cm2
  * Total area of all lesions bigger than 8cm2
  * Lesions other than on the femoral condyle and/or trochlea
  * Any evidence of the following diseases in the target joint: septic arthritis; inflammatory joint disease; gout; recurrent episodes of pseudogout; Paget disease of bone; ochronosis; acromegaly; hemochromatosis;Wilson disease; primary osteochondromatosis; heritable disorders; collagen gene mutations
  * Presence of a clinically relevant cartilage lesion on the patella (second lesion)
  * Patellofemoral cartilage lesion
  * Presence of relevant complex knee injuries affecting bone and/or ligaments
  * Osteochondritis dissecans: recent (within 1 year before baseline); depth of lesion >0.5 cm; subchondral sclerosis
  * Advanced osteoarthritis (as defined by Radiographic Atlas of Osteoarthritis, grade 2-3)
  * Varus or valgus malalignment exceeding 5° (kissing lesions out)
* Medical history:

  * gravidity (Pregnancy)
  * breast feeding
  * presence of multiple severe allergies (including porcine collagen, streptomycin and penicillin)
  * Osteoarthritis
  * Current diagnosis of osteomyelitis
  * Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
  * A blood result showing liver enzymes (serum glutamic oxaloacetic transaminase, serum glutamic pyruvic transaminase, alkaline phosphatase) of more than 2 times the upper limit of normal or any other result that in the clinical investigator's mind is clinically important
  * C-reactive protein level greater than 10 mg/L
  * Uncontrolled diabetes
  * Renal insufficiency
  * Previous pacemaker implantation
  * Any concomitant painful or disabling disease of the spine, hips, or lower limbs that would interfere with evaluation of the afflicted knee
  * Mosaicplasty (osteochondral autograft transfer system)
  * Microfracture performed less than 1 year before baseline
  * Received hyaluronic acid intra-articular injections into the afflicted knee within the last 6 months of baseline Meniscal transplant (previous/present)
  * Meniscal suture with meniscal arrows ipsilaterally (present or previous if not resorbed)
  * Taking specific osteoarthritis drugs, such as chondroitin sulfate, diacerein, n-glucosamine, piascledine, and capsaicin, within 2 weeks of the baseline visit
  * Corticosteroid therapy by systemic or intra-articular route within the last month of baseline or intramuscular or oral corticosteroids within the last 2 weeks of baseline
  * Chronic use of anticoagulants
  * Patients with human immunodeficiency virus, hepatitis, or syphilis
  * Malignancy
  * Alcohol and drug (medication) abuse
  * Poor general health condition as judged by investigator
  * Body mass index >35 kg/m2
  * Medication:chronic treatment with steroids or growth factors (immunomodulatory drugs)
* Other:

  * Participation in concurrent clinical trials
  * Participation in a previous clinical trial within 1 year

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
1-Safety for the patient | until 24 months
  Safety will be assessed by the incidence of adverse reactions and adverse events. Expected postoperative complications also occurring in the standard procedure are: pain, swelling and hematoma, casually post-anesthetic nausea, vomiting or fever.
2- Stability of the graft | until 24 months
  It will be assessed by Magnetic Resonance Imaging (MRI) technique at 6, 12 and 24 months indicating if the graft is in place and if there are signs of complications. Parameters to be evaluated are: filling of the defect, integration of the border zone to the adjacent cartilage, intactness of the subchondral lamina, intactness of the subchondral bone, and relative signal intensities of the repair tissue compared to the adjacent native cartilage.

SECONDARY OUTCOMES:
Subjective pain relief | until 24 months
  Subjective relief of pain for the patient will be assessed using the International Cartilage Repair Society (ICRS) Cartilage Injury Evaluation Package which includes the pre- and postsurgical evaluation of general medical conditions, pain, activity level as well as functional and morphological status.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Jakob, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Mumme M, Barbero A, Miot S, Wixmerten A, Feliciano S, Wolf F, Asnaghi AM, Baumhoer D, Bieri O, Kretzschmar M, Pagenstert G, Haug M, Schaefer DJ, Martin I, Jakob M. Nasal chondrocyte-based engineered autologous cartilage tissue for repair of articular cartilage defects: an observational first-in-human trial. Lancet. 2016 Oct 22;388(10055):1985-1994. doi: 10.1016/S0140-6736(16)31658-0. PMID 27789021